CLINICAL TRIAL: NCT03636178
Title: Three Dimensional Evaluation of Nasolabial Changes Following Classic Versus Modified Alar Base Suture After Le Fort I Osteotomy
Brief Title: 3D Evaluation of Nasolabial Changes Following Classic Versus Modified Alar Base Suture After Le Fort I Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samy, Oral and Maxillofacial surgeon, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-07-01
Record Dates: First submitted 2018-08-12; First posted 2018-08-17 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Le Fort; I
Keywords: alar base; le fort I osteotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st group (Other): 20 patients out of 40 will be enrolled into the study including males and females above 18 years old
  Interventions: Procedure: Classic alar base suture technique
- 2nd group (Other): 20 patients out of 40 will be enrolled in the study including males and females above 18 years old
  Interventions: Procedure: Modified alar base suture technique

INTERVENTIONS:
Procedure: Classic alar base suture technique — An index finger will be used to apply extraoral pressure on the alar base region, and a dentate forceps will grasp this tissue through the intraoral incision. A suture bite will be taken at this point through the tissue previously held by the forceps. The same procedure will be applied on the opposite side. After passing the suture on both sides, it will be tightened with attention to the alar base response. If the alar base suture will be judged to be adequate, the vestibular incision will then be closed in a routine fashion, with or without performing a V-Y lip closure
  Arms: 1st group
Procedure: Modified alar base suture technique — The alar base will be marked with 3 landmarks: left alar base (point LAB), columella (point C), and right alar base (point RAB). A needle will be inserted through the skin at the nasofacial skin fold and exited through the fibroareolar tissue. A nonabsorbable suture without a needle will be inserted through the needle from the oral cavity to the outside. The needle will be retracted through point RAB without leaving the skin point, then returned to the oral cavity in a medial position. Finally the needle will be retracted from point RAB, leaving the suture through the soft tissue. The same procedure will be repeated on the other side. The 2 free ends of the sutures will be then tied together after passing through a hole made in the nasal spine.
  Arms: 2nd group

SUMMARY:
Three dimensional evaluation of nasolabial changes following classic versus modified alar cinch suture after Le Fort I osteotomy using cone beam computed tomography

DETAILED DESCRIPTION:
Intra operative procedures: (For all groups) All surgical operations will be performed or supervised by one of the authors (MdK). Intraoperative antibiotics will be given(1000 mg cefazolin and 500 mg metronidazole). After nasotracheal intubation, the mucobuccal fold of the maxilla will be infiltrated with local anaesthetic (articaine ; Ultracain DS Forte). The Le Fort I procedure will be started with an incision in the gingivobuccal sulcus from the canine on the one side to the canine on the other side. After elevation of the mucoperiosteum and nasal mucosa, the osteotomy line will be designed with a fine burr, after which the cut will be made with a reciprocal saw. The lateral nasal walls and nasal septum will be osteotomized with a nasal osteotome. The piriform aperture and when necessary the nasal spine will be rounded off. After mobilization of the maxilla, it will be positioned in the planned position using an acrylic wafer. Fixation will be performed with four 1.5-mm miniplates, one paranasal and one on the buttress on each side. The mucosa will be closed with a 4-0 Vicryl suture (Ethicon ; Johnson and Johnson Medical, Norderstedt, Germany).

The alar cinch procedure will be performed through the intraoral incision as follows:

In the comparator ( control ) group:

The classic method of alar cinching will be performed in the following manner: An index finger will be used to apply extraoral pressure on the alar base region, and a dentate forceps will grasp this tissue through the intraoral incision. A suture bite will be taken at this point through the tissue previously held by the forceps. The same procedure will be applied on the opposite side. After passing the suture on both sides, it will be tightened with attention to the alar base response. If the alar base suture will be judged to be adequate, the vestibular incision will then be closed in a routine fashion, with or without performing a V-Y lip closure.

In the intervention group:

The alar base will be marked with 3 landmarks: the nasofacial skin fold at the left alar base (point LAB), the middle of the columella (point C), and the nasofacial skin fold at the right alar base (point RAB). A needle will be inserted through the skin at the nasofacial skin fold and exited through the fibroareolar tissue. A nonabsorbable suture without a needle will be inserted through the needle from the oral cavity to the outside. The needle will be retracted through point RAB without leaving the skin point, then returned to the oral cavity in a medial position. Finally the needle will be retracted from point RAB, leaving the suture through the soft tissue. The same procedure will be repeated on the other side. The 2 free ends of the sutures will be then tied together after passing through a hole made in the nasal spine.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with skeletal maxillomandibular deformity indicated for surgical correction by Le Fort I osteotomy.
2. Absence of clefts.
3. Absence of growth.
4. Patients must be willing for the surgical procedure and follow-up, with his informed consent.

Exclusion Criteria:

1. History of facial trauma with fractures of facial bones.
2. History of surgical operation in nasal region.
3. Facial asymmetry.
4. Patients with accompanying craniofacial syndromes.
5. Patients with any diseases that compromise bone or soft tissue healing.
6. Anterior open bite cases
7. Medically compromised patients not fit for general anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Widening of the alar base | 6 months postoperatively
  Postoperative increase in the alar base width in millimeters(mm) in comparison to the normal preoperative alar base width

SECONDARY OUTCOMES:
Nasal volume | 6 months postoperatively
  Postoperative increase or decrease in the nasal volume in cubic millimeters in comparison to the normal preoperative nasal volume

IPD SHARING:
Plan to Share IPD: No